CLINICAL TRIAL: NCT06418906
Title: The Relationships Between Equanimity, Mindfulness, and Self-Compassion, and Mental Health Outcomes
Status: Recruiting | Type: Observational
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Other Study IDs: 1005240113
Record Dates: First submitted 2024-05-13; First posted 2024-05-17 (Actual); Last update posted 2024-06-03 (Actual); Status verified 2024-05

CONDITIONS: Mindfulness; Mental Health Outcomes; Self-Compassion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Community adults aged 18 or above: This is a single-arm study with no intervention involved. Adults aged 18 or above from the community will be invited to fill out the same set of questionnaires on a total of two time points: baseline and two-week post-baseline.
  Interventions: Other: Self-reported questionnaires

INTERVENTIONS:
Other: Self-reported questionnaires — After participants agree to participate in this study, they will first fill out the set of questionnaires once. After two weeks, the research team will send them reminders to fill out the same set of questionnaires again.

SUMMARY:
This is an academic research study aiming to explore the relationships between equanimity, mindfulness, self-compassion, and mental health outcomes, and to examine the reliability and validity of the new measures in Hong Kong.

DETAILED DESCRIPTION:
The current research aims to validate two new measures, the Equanimity Scale (ES-16) and the Sussex-Oxford Compassion for the Self Scale (SOCS-S) in Hong Kong. Standard procedures of forward-backward translation of the ES-16 and SOCS-S were employed. Adults aged 18 or above will be recruited in the community to fill out a set of questionnaires two times on equanimity, mindfulness, self-compassion, and mental health outcomes (i.e., depression, anxiety, stress, wellbeing). Relationships between these variables will be explored. To assess test-retest reliability, participants will be invited to fill out the same set of questionnaires on a total of two time points: baseline and two-week post-baseline.

ELIGIBILITY:
Inclusion Criteria:

* aged 18 or above
* can read and type Chinese
* have means to access online surveys

No Exclusion Criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Community participants aged 18 or above
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-05 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Mindfulness (Five Facet Mindfulness Questionnaire - 20) | 2-week
  The 20-item Five Facet Mindfulness Questionnaire - 20 (FFMQ-20) will be used to measure mindfulness. Possible score range is 20 to 100, where higher scores indicate higher mindfulness.
Equanimity (Equanimity Scale) | 2-week
  The 16-item Equanimity Scale (ES-16) will be used to measure equanimity. Possible score range is 16 to 80, where higher scores indicate higher equanimity.
Self-compassion (Sussex-Oxford Compassion for the Self Scale) | 2-week
  The 20-item Sussex-Oxford Compassion for the Self Scale (SOCS-S) will be used to measure self-compassion. Possible score range is 20 to 100, where higher scores indicate higher self-compassion.
Depression (Patient Health Questionnaire - 9) | 2-week
  The nine-item Patient Health Questionnaire - 9 (PHQ-9) will be used to measure depression. Possible score range is 0 to 27, where higher scores mean more severe depression.
Anxiety (Generalized Anxiety Disorder - 7) | 2-week
  The seven-item Generalized Anxiety Disorder-7 (GAD-7) will be used to measure anxiety. Possible score range is 0 to 21, where higher scores indicate more severe anxiety.
Stress (Perceived Stress Scale - 10) | 2-week
  The 10-item Perceived Stress Scale - 10 (PSS) will be used to measure stress. Possible score range is 0 to 40, where higher scores indicate higher perceived stress.
Wellbeing (Short Warwick-Edinburgh Mental Wellbeing Scale) | 2-week
  The seven-item Short Warwick-Edinburgh Mental Wellbeing Scale (SWEMWBS) will be used to measure wellbeing. Possible score range is 0 to 35, where higher scores mean higher mental wellbeing.
Equanimity (Two-Factor Equanimity Scale) | 2-week
  The Two-Factor Equanimity Scale (EQUA-S) will be used to measure equanimity, for assessing convergent validity of the ES-16. Possible score range is 14 to 70, where higher scores indicate higher equanimity.
Self-compassion (Self-Compassion Scale - Short Form) | 2-week
  The 12-item Self-Compassion Scale - Short Form (SCS-SF) will be used to measure self-compassion, for assess convergent validity of the SOCS-S. Possible score range is 12 to 60, where higher scores indicate higher self-compassion.

SECONDARY OUTCOMES:
single-item measures on equanimity, mindfulness, self-compassion, depression, anxiety, stress (i.e., six items in total) | 2-week
  Six single-item exploratory weekly measures respectively measuring equanimity, mindfulness, self-compassion, depression, anxiety, stress. Possible score range for single-item measures on equanimity, mindfulness, self-compassion are 1 to 7, where higher scores indicate higher equanimity, mindfulness, self-compassion respectively. Possible score range for single-item measures on depression, anxiety are 0 to 3, where higher scores indicate more severe depression, anxiety respectively. Possible score range for single-item measure on stress is 0 to 4, where higher scores indicate higher perceived stress.

CONTACTS AND LOCATIONS:
Overall Officials: Hoi Chun Lok, MSocSc(CP), Principal Investigator — The University of Hong Kong
Locations (1):
- Department of Psychology, The University of Hong Kong, Hong Kong, Hong Kong